CLINICAL TRIAL: NCT03109912
Title: Do More, B'More, Live Fit: An Outpatient Fitness-training Pilot Program Designed to Optimize the Habit of Exercise in Adolescents and Young Adults With Cystic Fibrosis
Brief Title: Do More, B'More, Live Fit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00055571
Record Dates: First submitted 2017-02-22; First posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Cystic Fibrosis; Physical Activity
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): At the baseline fitness assessment, the FitBit daily step goal is set at the manufacturer standard 10,000 steps. Throughout the study, these 30 participants will receive generic, non-personalized encouragement and recommendations (if requested by the participant) for PA at routine clinic visits, baseline and follow-up assessments at 3 and 6 month clinic visits. At the 3-month and 6-month visits, exercise is reinforced with generic encouragement, export FitBit data and review any missing data concerning for equipment failure or user error.
- Exercise Intervention (Experimental): The baseline fitness assessment includes an additional 30-minutes for exercise prescriptions; participant FitBit daily step goal is set based on a collaborative review between the participant and PT and participants receive individualized exercise prescriptions based on their assessment. Throughout the study, these 30 participants will receive customized encouragement and personalized fitness recommendations for PA at routine visits, baseline and follow-up assessments at 3 and 6 month clinic visits. At the 3-month and 6-month visits, study team members meet again with the participant for an additional 30-45 minutes to reinforce exercise through exercise prescriptions and individualized encouragement, export FitBit data and review any missing data concerning for equipment failure or user error and address any specific exercise concerns. FitBit daily step goals may be adjusted based on collaborative review between the participant and PT.
  Interventions: Behavioral: Personalized-Coaching Interventions; Behavioral: Motivational Messages; Behavioral: Online Exercise Tutorials; Behavioral: Social Support and Peer Challenges

INTERVENTIONS:
Behavioral: Personalized-Coaching Interventions — At the baseline fitness assessment, participants receive exercise prescriptions based upon their individual assessment. One of the ultimate exercise prescription goals is to achieve 30-minutes of an endurance-style exercise 5 times/week which may vary depending upon baseline fitness assessment. Aside from team sports, endurance-style exercise prescriptions may include simply walking, jump roping or stair climbing to more complex Tabata-style workouts. Two additional physical therapy (PT) 30-minute appointments are scheduled about 4-6 weeks and 8-10 weeks from enrollment. These 30-minute PT follow-up appointments will vary based on initial assessment and previous exercise prescription success but will include strength training for major muscles groups and/or flexibility exercises with yoga as well as reinforcement of previously learned techniques. PT will add additional individualized recommendations.
  Arms: Exercise Intervention
Behavioral: Motivational Messages — Intervention participants are enrolled to receive motivational messages starting 14 days after enrollment via preferred contact method (SMS, telephone call and/or email) every 3-4 days over the 6-month study period.
  Arms: Exercise Intervention
Behavioral: Online Exercise Tutorials — Participants are given access to Do More, B'More, Live Fit webpage which includes spotlighted exercises, instructional exercise photos and videos.
  Arms: Exercise Intervention
Behavioral: Social Support and Peer Challenges — Participants are invited to join the Do More, B'More, Live Fit Activity Group via the FitBit Dashboard and are invited to friend the study team members and other exercise-intervention participants in order to take part in FitBit step-goal challenges.
  Arms: Exercise Intervention

SUMMARY:
Physical activity (PA) in individuals with cystic fibrosis (CF) improves exercise capacity, slows decline in lung function, increases mucus clearance and improves health-related quality of life (HRQoL). Establishing and maintaining an exercise routine remains challenging and programs promoting PA in people with CF have poor participation. Moreover, while the positive effects of physical conditioning on lung function have been well reported, conventional measurements of lung function may lack the sensitivity to reveal improvement in mild lung disease.

This randomized control trial (RCT; N = 60) evaluates the Do More, B'More, Live Fit, a 6-month fitness program designed to optimize exercise habits of 12-21 year-olds with CF through structured exercises with personalized coaching, exercise equipment including the FitBit Flex, online support and motivational messages delivered electronically. The intervention incorporates fitness preferences and encompasses endurance, strength and flexibility exercises while adjusting to physical fitness needs. The hypothesis is that intervention participants will have increased and sustained engagement and better health outcomes compared to control group participants. The investigators' specific aims are to:

1. Increase daily PA and measures of fitness
2. Improve lung clearance index (LCI) and participant HRQoL
3. Demonstrate feasibility, accessibility and satisfaction of intervention using semi-structured interviews

The results of this pilot evaluation of the Do More, B'More, Live Fit program will offer novel insight into factors that sustain engagement in exercise programs and identify if LCI is an appropriate clinical outcome to assess PA interventions. Results will inform future RCT of interventions to optimize exercise habits of adolescents with CF.

ELIGIBILITY:
Inclusion Criteria:

* 12-21 year-old patients with a diagnosis of cystic fibrosis that are cared for at Johns Hopkins
* Participants must have smart phone and/or computer with universal serial bus (USB) access to set-up FitBit Flex

Exclusion Criteria:

* Forced expiratory volume in 1 second (FEV1) < 40% predicted
* Individuals already participating in vigorous physical activity as assessed by the study team such as participating in year-round organized sports and/or aerobic exercise >30 minutes more than 5 times/week may or may not be included in this study at the discretion of the PI and study team.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2015-06-17 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Pulmonary function testing (Lung clearance index: LCI 2.5 and LCI 5.0) | Change from baseline at 6-months
  LCI is measured via multiple breath washout (MBW) using a device called the EXHALYZER D. MBW is a non-invasive test that measures how difficult it is for air to leave the lungs and currently, the use of the EXHALYZER D is investigational. For MBW, participants breathe oxygen for about 3-5 minutes using a mouthpiece and normal breathing without any special breathing maneuvers.
Daily activity via FitBit Step Count | Change from baseline at 6-months
  Daily step count (mean, median and highest daily) recorded through participant FitBit flex

SECONDARY OUTCOMES:
Pulmonary function testing (FEV1) | Change from baseline at 6-months
  Spirometry is obtained for FEV1 percent predicted
Self-reported daily activity via the Habitual Activity Estimation Scale (HAES) | Change from baseline at 6-months
  Self-reported activity will be measured via the HAES. The HAES is a questionnaire that measures self-reported light, moderate or strenuous activity for weekday and weekend activities. The HAES is a reliable and valid instrument in the pediatric and adult CF patient populations. Habitual activity will be recorded as a percentage of time when the participant was awake and performing light, moderate, and vigorous aerobic physical activity, strengthening and/or stretching exercises.
Health-related Quality of Life (HRQoL) via Cystic Fibrosis Questionnaire- Revised (CFQ-R) | Change from baseline at 6-months
  The CFQ-R, a HRQoL measure for people with CF that measures symptoms and treatment burden. It is a validated instrument for CF patients that scores QoL in 12 general domains, will be administered to assess the participant's HRQoL at baseline and 6-months from intervention onset. Scores for each domain will be expressed on a scale of 0-100.
Exercise capacity via Modified Shuttle Walk Test (MSWT) | Change from baseline at 6-months
  For the MSWT, participants are asked to walk 10-meter sets at a faster and faster speed until they are unable to continue to keep up with the increased speed or have symptoms including fatigue, dyspnea, chest pain that prevent them from continuing. It is a validated field test of exercise capacity in pediatric CF patients in which the participant walks shuttles of 10-meters in length at a progressively increasing pace. The number of shuttles completed will be recorded at baseline and 6-months from enrollment. Comparisons will be made between cohorts and between participant change from baseline to study conclusion at 6-months.
Semi-structured interview | Change from baseline at 6-months
  30-minute survey at follow-up 6-month appointments to assess acceptability and feasibility of the exercise interventions. Conducted by study team members with the participant and parent together, the one-time survey includes themes on intervention burden, benefits and/or concerns with interventions, willingness to continue interventions, suggestions to make interventions more feasible for regular use, perception of behavior change and technical challenges with interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Mogayzel, MD, Principal Investigator — Johns Hopkins University